CLINICAL TRIAL: NCT01005719
Title: Randomized, Crossover, Pharmacodynamic Study Comparing the Effects of Two Proton Pump Inhibitors
Brief Title: Study to Compare Gastric Inhibition of Two Proton Pump Inhibitors (CL2008-18)(P07815)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18135; CL2008-18; P07815 (Other: Merck)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2011-01-28 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Human Experimentation
MeSH Terms: interventions — omeprazole, sodium bicarbonate drug combination; Omeprazole; Sodium Bicarbonate; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zegerid (Experimental): Participants receiving Zegerid (omeprazole/sodium bicarbonate) in Periods 1, 2 or 3. All participants were randomized to a 3-way crossover design and received Zegerid Capsules (20 mg omeprazole/ 1100 mg sodium bicarbonate), Prevacid Capsules (15 mg lansoprazole), or no treatment in a random order. All participants also took approximately 2 oz of water with their medication.
  Interventions: Drug: Zegerid
- Prevacid® (Active Comparator): Participants receiving Prevacid® (lansoprazole) in Periods 1, 2 or 3. All participants were randomized to a 3-way crossover design and received Zegerid Capsules (20 mg omeprazole/ 1100 mg sodium bicarbonate), Prevacid Capsules (15 mg lansoprazole), or no treatment in a random order. All participants also took approximately 2 oz of water with their medication.
  Interventions: Drug: Prevacid®
- No treatment (No Intervention): Participants receiving No treatment in Periods 1, 2 or 3. All participants were randomized to a 3-way crossover design and received Zegerid Capsules (20 mg omeprazole/ 1100 mg sodium bicarbonate), Prevacid Capsules (15 mg lansoprazole), or no treatment in a random order. All participants took approximately 2 oz of water once daily for 7 days.

INTERVENTIONS:
Drug: Zegerid — Zegerid (20 mg omeprazole/ 1100 mg sodium bicarbonate) taken with approximately 2 oz of water once daily for 7 days.
  Other Names: omeprazole/sodium bicarbonate, SCH 900934
  Arms: Zegerid
Drug: Prevacid® — Prevacid (15 mg lansoprazole) taken with approximately 2 oz of water once daily for 7 days.
  Other Names: lansoprazole
  Arms: Prevacid®

SUMMARY:
This study will determine differences between Proton Pump Inhibitors (PPI) formulations relative to their effects on gastric acidity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-Asian, male or non-lactating, non-pregnant female participants who are 18-65 years of age.
* Clinical laboratory test must be within normal limits or clinically acceptable to the Investigator/Sponsor.
* Participants must have normal or clinically acceptable physical exam and ECG.
* Participants must be free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations, procedures, or participation.
* Able to understand and comply with study procedures required and able and willing to provide written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* History of hypersensitivity, allergy or intolerance to omeprazole, or other proton pump inhibitors
* History of peptic ulcer disease or other acid related gastrointestinal symptoms or heartburn with a frequency of more than one/month.
* Positive H. pylori breath test at screening.
* Participation in any study of an investigational treatment in the 30 days before Screening or participation in another study at any time during the period of this study
* Any significant medical illness that would contraindicate participation in the study
* Gastrointestinal disorder or surgery leading to impaired drug absorption
* Any significant mental illness, such as schizophrenia or bipolar disorder
* History (in the past year) suggestive of alcohol or drug abuse or dependence, or excessive alcohol use (>2 units per day on average; for example >2 bottles of beer, >2 glasses of wine, >2 ounces of liquor/spirits), or excessive alcohol use during the study
* Any abnormal Screening laboratory value that is clinically significant in the investigator's opinion
* Currently using or use of any prescription or over the counter (OTC) medications that affect gastrointestinal function, including first generation antihistamines (e.g. diphenhydramine) and anticholinergic agents within 7 days prior to 1st treatment administration.
* Currently using, or use within 14 days of first treatment administration, or having a history of frequent use of antacids, OTC or Prescription (Rx) H2 receptor antagonists, or OTC or Rx use of proton pump inhibitors.
* Positive urine drug/alcohol test at Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Zegerid-Prevacid®-No Treatment: Participants received Zegerid in Period 1, Prevacid® in Period 2 and No treatment in Period 3.
- Zegerid-No Treatment-Prevacid®: Participants received Zegerid in Period 1, No treatment in Period 2 and Prevacid® in Period 3
- Prevacid®-Zegerid-No Treatment: Participants received Prevacid® in Period 1, Zegerid in Period 2 and No treatment in Period 3
- Prevacid®-No Treatment-Zegerid: Participants received Prevacid® in Period 1, No treatment in Period 2 and Zegerid in Period 3
- No Treatment-Zegerid-Prevacid®: Participants received No treatment in Period 1, Zegerid in Period 2 and Prevacid® in Period 3
- No Treatment-Prevacid®-Zegerid: Participants received No treatment in Period 1, Prevacid® in Period 2 and Zegerid in Period 3
Period: Period 1
Arm/Group | Zegerid-Prevacid®-No Treatment | Zegerid-No Treatment-Prevacid® | Prevacid®-Zegerid-No Treatment | Prevacid®-No Treatment-Zegerid | No Treatment-Zegerid-Prevacid® | No Treatment-Prevacid®-Zegerid
Started | 10 | 10 | 10 | 11 | 11 | 11
Completed | 10 | 10 | 10 | 10 | 11 | 10
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Delay in completing study procedures | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Zegerid-Prevacid®-No Treatment | Zegerid-No Treatment-Prevacid® | Prevacid®-Zegerid-No Treatment | Prevacid®-No Treatment-Zegerid | No Treatment-Zegerid-Prevacid® | No Treatment-Prevacid®-Zegerid
Started | 10 | 10 | 10 | 10 | 11 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1
Period: Period 3
Arm/Group | Zegerid-Prevacid®-No Treatment | Zegerid-No Treatment-Prevacid® | Prevacid®-Zegerid-No Treatment | Prevacid®-No Treatment-Zegerid | No Treatment-Zegerid-Prevacid® | No Treatment-Prevacid®-Zegerid
Started | 10 | 10 | 10 | 10 | 10 | 9
Completed | 10 | 10 | 10 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Sustained Difference in Inhibition of Intragastric Acidity Based on Median pH Values Between the Two Active Study Treatments at Steady-state on Day 7
Description: Median intragastric pH scores were collected at 5 minute intervals after treatment dose. The achievement of sustained difference was the earliest time for which a statistically significant difference was observed in the median intragastric pH scores for 3 consecutive 5-minute intervals. The earliest 3 time points for which a statistically significant difference was observed between the median intragastric pH values for the two active treatments for three consecutive 5-minute intervals are shown here.
Time Frame: Treatment dose to 4-hr post-dose on Day 7
Population: Participants who received at least one dose of study treatment, and did not have missing values.
Measure: Median (Full Range); unit: pH
Groups:
- Zegerid: Participants receiving Zegerid in Periods 1, 2 or 3.
  All participants were randomized to a 3-way crossover design and received Zegerid Capsules (20 mg omeprazole/ 1100 mg sodium bicarbonate), Prevacid Capsules (15 mg lansoprazole), or no treatment in a random order.
- Prevacid®: Participants receiving Prevacid® in Periods 1, 2 or 3.
  All participants were randomized to a 3-way crossover design and received Zegerid Capsules (20 mg omeprazole/ 1100 mg sodium bicarbonate), Prevacid Capsules (15 mg lansoprazole), or no treatment in a random order.
Arm/Group | Zegerid | Prevacid®
Number analyzed (Participants) | 59 | 59
pH
  10-15 Minutes Post-dose on Day 7 | 2.600 [0.52 to 7.94] | 1.820 [0.64 to 6.38]
  15-20 Minutes Post-dose on Day 7 | 3.230 [0.45 to 8.16] | 1.760 [0.59 to 6.78]
  20-25 Minutes Post-dose on Day 7 | 4.920 [0.34 to 8.25] | 1.950 [0.45 to 7.04]
Statistical Analysis 1: Comparison: Zegerid vs Prevacid®; Test type: Superiority or Other; p = 0.0242, Wilcoxon (Mann-Whitney) — p-value for 10-15 mins Post-dose on Day 7. No adjustments were made for multiple comparisons. P-values <= 0.05 were reported as statistically significant
Statistical Analysis 2: Comparison: Zegerid vs Prevacid®; Test type: Superiority or Other; p = 0.0270, Wilcoxon (Mann-Whitney) — p-value for 15-20 mins Post-dose on Day 7. No adjustments were made for multiple comparisons. P-values <= 0.05 were reported as statistically significant
Statistical Analysis 3: Comparison: Zegerid vs Prevacid®; Test type: Superiority or Other; p = 0.0067, Wilcoxon (Mann-Whitney) — p-value for 20-25 mins Post-dose on Day 7. No adjustments were made for multiple comparisons. P-values <= 0.05 were reported as statistically significant

2. Secondary Outcome: Achievement of Sustained Difference in Inhibition of Intragastric Acidity Based on Median pH Values Between the Two Active Study Treatments at Steady-state on Day 1
Description: as for outcome 1
Time Frame: Treatment dose to 4-hr post-dose on Day 1
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: pH
Arm/Group | Zegerid | Prevacid®
Number analyzed (Participants) | 59 | 57
pH
  10-15 Minutes Post-dose on Day 1 | 1.330 [0.28 to 8.81] | 1.070 [0.23 to 6.37]
  15-20 Minutes Post-dose on Day 1 | 1.420 [0.19 to 8.40] | 1.080 [0.27 to 2.90]
  20-25 Minutes Post-dose on Day 1 | 1.590 [0.15 to 9.00] | 0.990 [0.10 to 4.67]
Statistical Analysis 1: Comparison: Zegerid vs Prevacid®; Test type: Superiority or Other; p = 0.0465, Wilcoxon (Mann-Whitney) — p-value for 10-15 mins Post-dose on Day 1
Statistical Analysis 2: Comparison: Zegerid vs Prevacid®; Test type: Superiority or Other; p = 0.0012, Wilcoxon (Mann-Whitney) — p-value for 15-20 mins Post-dose on Day 1
Statistical Analysis 3: Comparison: Zegerid vs Prevacid®; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — p-value for 20-25 mins Post-dose on Day 1

3. Secondary Outcome: The Difference in the Onset of Action Based on Median pH Values Between the Two Active Treatments Compared to No Treatment on Day 1 and Day 7
Description: Median intragastric pH scores were collected at 5 minute intervals after treatment dose. The difference in the onset of action was the earliest 5 minute interval (from start of interval to end of interval) for which each active treatment presented a statistically significantly advantage over No treatment based on median pH values. The earliest 5 minute interval showing the difference in onset of action is reported here.
Time Frame: Treatment dose to 4-hr post-dose on Day 1 and Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: pH
Groups:
- No Treatment: Participants receiving No treatment in Periods 1, 2 or 3.
  All participants were randomized to a 3-way crossover design and received Zegerid Capsules (20 mg omeprazole/ 1100 mg sodium bicarbonate), Prevacid Capsules (15 mg lansoprazole), or no treatment in a random order.
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
pH
  Day 1 (0-5 mins), (N=59, N=57, N=59) | 1.050 [0.37 to 6.83] | 1.180 [0.27 to 7.03] | 0.92 [0.10 to 4.01]
  Day 7 (0-5 mins), (N=59, N=59, N=59) | 1.840 [0.10 to 6.78] | 1.950 [0.50 to 7.88] | 0.82 [0.25 to 7.00]
Statistical Analysis 1: Comparison: Zegerid vs No Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — The statistical analysis is for Day 1 (0-5 mins)
Statistical Analysis 2: Comparison: Prevacid® vs No Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — The statistical analysis is for Day 1 (0-5 mins)
Statistical Analysis 3: Comparison: Zegerid vs No Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — The statistical analysis is for Day 7 (0-5 mins)
Statistical Analysis 4: Comparison: Prevacid® vs No Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — The statistical analysis is for Day 7 (0-5 mins)

4. Secondary Outcome: Median Time to Achieve Intragastric pH > = 3.5 for a 10-Minute Period
Description: The time required to achieve an intragastric pH ≥3.5 that is reached for 10 consecutive minutes after drug administration on the 1st and 7th days of dosing.
Time Frame: Treatment dose to 4-hr post-dose on Day 1 and Day 7
Population: Participants who received at least one dose of study treatment, and did not have missing values.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
Minutes
  Day 1 (N=59, N=57, N=59) | 64.867 [0.00 to 240.00] | 108.867 [0.00 to 240.00] | 240.00 [2.27 to 240.00]
  Day 7 (N=59, N=59, N=59) | 22.667 [0.00 to 240.00] | 66.667 [0.00 to 240.00] | 240.00 [0.00 to 240.00]

5. Secondary Outcome: Percentage Time Intragastric pH >4 During the First 4 Hours After Dosing on Day 7
Time Frame: Treatment dose to 4 hours Post-dose on Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Percentage of time
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
Percentage of time | 64.639 [1.36 to 100.00] | 44.194 [0.00 to 100.00] | 6.056 [0.00 to 70.28]

6. Secondary Outcome: Median 24-hr Intragastric pH on Day 7
Description: The median intragastric pH values were recorded over a 24-hr period.
Time Frame: Treatment dose to 24-hour post-dose on Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: pH
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
pH | 3.600 [0.69 to 6.64] | 3.100 [0.22 to 6.58] | 0.800 [0.10 to 3.19]

7. Secondary Outcome: Percentage of Time Intragastric is pH >4 Over 24-hour Period on Day 7
Time Frame: Treatment dose to 24-hour post-dose on Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Percentage of time
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
Percentage of time | 40.538 [1.39 to 81.26] | 36.917 [1.18 to 92.75] | 4.852 [0.26 to 35.28]

8. Secondary Outcome: Percentage of Time Intragastric pH >3.5 Over 24-hour Period on Day 7
Time Frame: Treatment dose to 24-hours post-dose on Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Percentage of Time
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
Percentage of Time | 51.321 [1.81 to 89.27] | 43.990 [3.40 to 93.44] | 7.927 [0.34 to 41.15]

9. Secondary Outcome: Number of Participants With Intragastric pH >4 for More Than 50% of the Time on Day 7
Description: Number of participants maintaining intragastric pH > 4 for at least 12 hrs at
  steady-state on Day 7
Time Frame: Treatment dose to 24-hour post-dose on Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Number; unit: Participants
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
Participants | 26 | 18 | 0

10. Secondary Outcome: Number of Participants With Intragastric pH >3.5 for More Than 50% of the Time on Day 7
Description: Number of participants maintaining intragastric pH > 3.5 for at least 12 hrs at
  steady-state on Day 7
Time Frame: Treatment dose to 24-hour post-dose on Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Number; unit: Participants
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
Participants | 30 | 23 | 0

11. Secondary Outcome: Percentage of Time Intragastric pH >4 Over the Nocturnal Period on Day 7
Time Frame: Treatment dose to 24-hour post-dose on Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Percentage of Time
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 58 | 58
Percentage of Time | 9.236 (17.426) [0.00 to 65.28] | 9.685 (17.008) [0.00 to 90.24] | 0.028 [0.00 to 61.01]

12. Secondary Outcome: Time to Achieve Sustained Intragastric pH > 3.5 at Steady-state on Day 7
Description: The first time to sustain median pH > 3.5 for at least 3 successive 5-minute periods within the first 2 hours after dosing with Zegerid Capsules, and Prevacid Capsules, or No treatment on the 7th day of respective treatments. If this condition was not met for any time point within the first 2 hours following dosing, a score of 120 minutes was imputed.
Time Frame: Treatment dose to 2-hours post-dose on Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 59 | 59
Minutes | 25.000 [5.00 to 120.00] | 65.000 [5.00 to 120.00] | 100.000 [5.00 to 120.00]

13. Secondary Outcome: Time to Onset of Inhibition of Acid Secretion on Day 1
Description: The onset of inhibition of acid secretion was the first time to sustain median pH >3.5 for each of the twenty-four successive 5-minute periods. If this condition was not met for any time point within the first 4 hours following dosing, a score of 240 minutes was imputed.
Time Frame: Treatment dose to onset of event on Day 1
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 57 | 59
Minutes | 240.00 (71.663) [5.00 to 240.00] | 240.00 (48.209) [80.00 to 240.00] | 240.00 (18.226) [100.00 to 240.00]

14. Secondary Outcome: Number of Participants Maintaining Intragastric pH > 4 for at Least 12 Hours on Day 1
Time Frame: Treatment dose to 24-hr post-dose on Day 1
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Number; unit: Participants
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 57 | 59
Participants | 8 | 5 | 0

15. Secondary Outcome: Number of Participants Maintaining Intragastric pH > 3.5 for at Least 12 Hours on Day 1
Time Frame: Treatment dose to 24-hr post-dose on Day 1
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Number; unit: Participants
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 57 | 59
Participants | 11 | 11 | 0

16. Secondary Outcome: Percentage of Time Intragastric pH >4 Over the Nocturnal Period on Day 1
Time Frame: Treatment dose to 24-hour post-dose on Day 1
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Percentage of Time
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 57 | 59
Percentage of Time | 0.681 [0.00 to 65.15] | 1.987 [0.00 to 98.68] | 0.111 [0.00 to 36.49]

17. Secondary Outcome: Percentage of Time Intragastric pH >4 During the First 4 Hours on Day 1
Time Frame: Treatment dose to 4-hours post-dose on Day 1
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Percentage of Time
Arm/Group | Zegerid | Prevacid® | No Treatment
Number analyzed (Participants) | 59 | 57 | 59
Percentage of Time | 21.500 [0.00 to 91.22] | 9.525 [0.00 to 73.26] | 3.667 [0.00 to 58.64]

18. Secondary Outcome: Time to Achieve Sustained Advantage Over No Treatment During the First 4 Hours After Dosing
Description: The earliest time during the first 4 hours after dosing that the median
  pH for the treatment is over 1 unit higher than that for the No treatment during the next three 5 minute intervals. (When this condition does not occur, the time to sustained advantage will be imputed as 4 hours.)
Time Frame: Treatment dose to event on Day 1 and Day 7
Population: Participants who received at least one dose of a study treatment, and presented valid data from all three study periods.
Measure: Median (Full Range); unit: Minutes
Groups:
- Prevacid®: Participants receiving in Prevacid® Periods 1, 2 or 3.
  All participants were randomized to a 3-way crossover design and received Zegerid Capsules (20 mg omeprazole/ 1100 mg sodium bicarbonate), Prevacid Capsules (15 mg lansoprazole), or no treatment in a random order.
Arm/Group | Zegerid | Prevacid®
Number analyzed (Participants) | 59 | 59
Minutes
  Day 1 (N=59, N=57) | 35.000 [0 to 240] | 85.000 [0 to 240]
  Day 7 (N=59, N=59) | 10.000 [0 to 240] | 5.000 [0 to 240]

ADVERSE EVENTS:
Description: Adverse events were collected for all participants who received at least one dose of study treatment.
Arm/Group | Zegerid | Prevacid® | No Treatment
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/61 | 0/62
Other Adverse Events (participants affected / at risk) | 4/60 | 8/61 | 5/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zegerid (N=60) | Prevacid® (N=61) | No Treatment (N=62)
Appendicitis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zegerid (N=60) | Prevacid® (N=61) | No Treatment (N=62)
Headache (Nervous system disorders) | 2 | 4 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other